CLINICAL TRIAL: NCT06914765
Title: A Pilot Study Evaluating the Safety and Efficacy of Endoscopic Sleeve Gastroplasty (ESG) in Obese Adolescents
Brief Title: ESG in Obese Adolescents
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Michael Manfredi, Attending Physician, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-021643
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Obese Adolescents; Obesity, Morbid; Obesity/Therapy
Keywords: Obesity; Pediatrics; Adolescents; BMI ≥95th percentile; Weight Loss; Weight Management; Endoscopic Sleeve Gastroplasty; Bariatric Procedure
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ESG Intervention (Experimental)
  Interventions: Device: Endoscopic Sleeve Gastroplasty (ESG) Procedure

INTERVENTIONS:
Device: Endoscopic Sleeve Gastroplasty (ESG) Procedure — The ESG procedure will be performed under general anesthesia monitored by an anesthesiologist. The device that will be used is called the Apollo Endosurgery ESG System, which is the only FDA approved device for the reduction of stomach volume through endoscopic sleeve gastroplasty for adult patients with obesity. This device works by being attached to a standard upper endoscope and is inserted through the mouth and goes into the stomach. When in the stomach, the back and front wall of the stomach will be stitched together to reduce the size of the stomach and help decrease the amount of food a patient can eat and drink at one time before feeling full.

SUMMARY:
The primary goal of this pilot study is to learn if the use of the Apollo Endosurgery ESG System is a safe, well tolerated intervention for weight loss in adolescents with obesity.

Secondary outcomes will evaluate the effectiveness of Endoscopic Sleeve Gastroplasty (ESG) in long-term reduction of weight, improvements in obesity-related co-morbidities and improvements in quality of life.

Participants will:

* Have their stomach volume reduced with the ESG procedure (study intervention), rather than with a bariatric surgery, under general anesthesia
* Undergo pregnancy testing (female participants only)
* Be admitted overnight to the hospital for recovery and monitoring following the ESG procedure
* Have a physical examination performed at study follow-up visits
* Participate in surveys about any side effects from the procedure and about quality of life
* Follow-up with the study team.
* Participants will still be seen in the multidisciplinary Bariatrics Clinic team consisting of an obesity medicine doctor, registered dietician, physical activity specialist, and psychologist as part of normal standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, age ≥ 12 years and ≤17 years at the time of study initiation (defined as the time of consent for participation in the pilot study).
2. BMI ≥95th percentile to 120% of the 95th percentile on the Centers for Disease Control and Prevention (CDC) growth curve with at least one obesity related comorbidity; OR BMI ≥ 120% of the 95th percentile on the CDC growth curve regardless of the presence or absence of comorbidities. Clinically significant obesity related comorbidities including type 2 diabetes mellitus, idiopathic intracranial hypertension (IIH), non-alcoholic steatohepatitis (NASH) now called metabolic dysfunction-associated steatohepatitis (MASH), Blount's disease, Slipped Capital Femoral Epiphysis (SCFE), sleep apnea defined as AHI ≥ 5, Gastroesophageal Reflux Disease (GERD), hypertension, or dyslipidemia.
3. Must have a documented history of weight management and weight loss attempts with supervised diets and exercise programs for at least 6 months from a Healthy Weight provider.
4. All female subjects must have a negative serum pregnancy test.
5. Has a signed note from a medically supervised weight loss program that the patient demonstrates commitment to nutrition, psychological, and physical activity evaluations and follow-ups in the Healthy Weight clinics, without frequent non-compliance or no-shows.
6. Demonstrates ability to understand what dietary and physical activity changes will be required for optimal postoperative outcomes based on psychology assessment.
7. Evidence for mature decision making, with appropriate understanding of potential risks and benefits of the procedure as deemed by a clinical psychologist.
8. No documented genetic cause for obesity or excessive weight gain such as Prader-Willi syndrome
9. Evidence that family and patient have the ability and motivation to comply with recommended treatments pre- and postoperatively. Evidence may include a history of reliable attendance at office visits for weight management and compliance with other medical needs.
10. Female participants must agree to avoid pregnancy for the duration of the study and acknowledge that they will be withdrawn from the study if they do become pregnant.
11. Patients agree to refrain from any type of additional weight loss surgery, reconstructive surgery, or weight-altering medications that would affect body weight.
12. Signed consent form from parent or guardian and signed assent for un-emancipated minors.

Exclusion Criteria:

1. Previous interventional/surgical treatment of obesity or prior gastric surgery.
2. Females who are pregnant or lactating.
3. Uncontrolled hypothyroidism or adrenal related obesity as determined by the investigator.
4. Known congenital or acquired anomalies of the GI tract such as esophageal or cricopharyngeal narrowing or stricture; distorted esophagus, esophageal pouch or pyloric stenosis.
5. Severe cardiovascular, cerebrovascular and/or cardiopulmonary disease or other serious organic disease that makes the subject a high-risk candidate as determined by the investigator.
6. Chronic or acute upper gastrointestinal bleeding conditions, e.g. gastric or esophageal varices; or esophageal or gastric disorders including uncontrolled diarrhea, dysmotility, or Barrett's Esophagus.
7. History of malignant hyperthermia, having a prior allergic reaction to general anesthesia, having a known difficult airway, or if the patient is not a candidate for general anesthesia.
8. Immunocompromised status such as that resulting from chronic oral steroid use, chemotherapeutic agents, or immune deficiency disorders or history or presence of pre-existing autoimmune connective tissue disease, i.e., systemic lupus erythematosus or scleroderma as determined by the treating investigator.
9. Subjects with uncontrolled psychiatric conditions including eating disorders (e.g., bulimia, binge eating disorder) as defined in the Diagnostic and Statistical Manual of Mental Disorders (DSM) 5
10. Acute or chronic infections (localized or systemic);
11. Significant movement limitations of lower extremities (e.g., cannot walk without the use of, or assistance from, a brace, cane, crutch, another person, prosthetic device, wheelchair, or other assistive device or is severely limited in their ability to walk due to an arthritic, neurological, or orthopedic condition).
12. Recently (within previous 3 months) prescribed or initiated therapy with medication(s) known to cause significant weight gain or weight loss including but not limited to a glucagon-like peptide-1 (GLP-1) Receptor Agonist, or is likely to require treatment with such medication(s) during the study.
13. Currently taking or has taken within the previous 3-months prescription or over-the-counter weight loss medications (e.g., medications and/or supplements containing ephedrine, phenylpropanolamine, amphetamines, etc.). Additionally, the subject must agree to refrain from use of such medications and weight loss/appetite suppressing dietary supplements during the course of the trial including the subject eligibility assessment period;
14. Weight loss of at least 5kg within the previous 3 months;
15. Patient with documented medical history/diagnosis of a mood disorder including, but not limited to active substance abuse, a history of psychoses, uncontrolled depression, suicidal attempts or current suicidal tendencies or ideations; or documented history of drug and/or alcohol abuse within one year of the screening visit;
16. The participant is currently enrolled in another investigational drug or device trial that has not completed the primary endpoint or that clinically interferes with this study.
17. Current cigarette smokers, vaping, alcohol, or marijuana use.
18. Patients with connective tissue disorders
19. Subjects in whom endoscopic surveillance of the stomach may be required including but not limited to Crohn's disease, Ulcerative Colitis, personal or family history of familial and non-familial adenomatous syndromes, or Lynch syndrome;
20. Conditions that, in the opinion of the investigator, may jeopardize the subject's well-being and/or the soundness of this clinical study.

At time of the ESG procedure, if the PI sees any evidence of the following: Hiatal hernia >2 cm, esophageal or gastric varices, ulcers of the stomach and or duodenum, esophageal or duodenal stenosis, or gastric or duodenal polyps, or Gastric Antral Vascular Ectasia.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Determine whether use of the Apollo Endosurgery ESG System is a safe, well tolerated intervention for weight loss in our study population | 24 months
  Number of procedure related adverse events will be collected. Severity of adverse events will be defined using the Clavien-Dindo Classification of Surgical Complications.

SECONDARY OUTCOMES:
Evaluate the effectiveness of ESG in long-term reduction of weight (BMI) | 24 months
  The primary parameter for assessing this objective will be a function of the percent change in BMI.
Evaluate the effectiveness of ESG in long-term reduction of weight (waist circumference) | 24 months
  Change in waist circumference, measured in centimeters.
Evaluate the effectiveness of ESG in long-term reduction of weight (obesity class) | 24 months
  Number of subjects who shift in class of obesity (class 3, class 2, and class 1).
Evaluate the impact of weight loss from ESG procedure on Type 2 Diabetes (with unchanged medication use) | 24 months
  Number of patients who show improvement in glycemic control parameters (fasting glucose, fasting insulin and HbA1c)
Evaluate the impact of weight loss from ESG procedure on Type 2 Diabetes (with decreased medication use) | 24 months
  Number of patients who show improvement in glycemic control parameters (fasting glucose, fasting insulin and HbA1c )
Evaluate the impact of weight loss from ESG procedure on Type 2 Diabetes (with medication discontinuation) | 24 months
  Number of patients who show improvement in glycemic control parameters (fasting glucose, fasting insulin and HbA1c)
Evaluate the impact of weight loss on obesity-related co-morbidities (reducing hypertension medication) | 24 months
  Number of subjects with a reduction in anti-hypertensive medication intake with no increase in blood pressure
Evaluate the impact of weight loss on obesity-related co-morbidities (reducing blood pressure) | 24 months
  Number of subjects with a reduction in blood pressure of 10/5mmHg with no increase in medication
Evaluate the impact of weight loss on obesity-related co-morbidities (stage of hypertension) | 24 months
  Number of subjects who show reduction in stage of hypertension (examples include Stage 2 Hypertension to Stage 1 Hypertension or Stage 1 Hypertension to no hypertension)
Evaluate the impact of weight loss on obesity-related co-morbidities (Dyslipidemia) | 24 months
  Number of subjects with decrease in low-density lipoprotein (LDL) by 10 mg/dL (with no increase in medication)
Evaluate the impact of weight loss on obesity-related co-morbidities (Dyslipidemia medications) | 24 months
  Number of subjects with reduction in medication intake with no adverse change in dyslipidemia indexes (LDL, TCL/HDL cholesterol ratio)
Evaluate the impact of weight loss on obesity-related co-morbidities (triglycerides) | 24 months
  Number of subjects with a decrease in fasting triglyceride to <150 mg/dL
Evaluate changes in hunger and satiety | 24-months
  Changes will be measured using a 2-item hunger-satiety questionnaire. This is a 2 item, self-report, measure that will assesses the subjects' hunger and fullness before and post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Manfredi, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size and sole location making study participation potentially identifiable for subjects, we do not plan to make IPD publicly available to other researchers. However, some data may be shared with research collaborators in the future upon obtaining Institutional Review Board approval and subject consent.